CLINICAL TRIAL: NCT04971486
Title: Effects of Feedback on Learning of a Motor Sequence Task and Resting State Connectivity
Brief Title: Feedback, Motor Sequence Learning, and Brain Connectivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Jill Stewart, PT, PhD, Associate Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Pro00097070
Record Dates: First submitted 2021-07-20; First posted 2021-07-21 (Actual); Last update posted 2022-01-13 (Actual); Status verified 2022-01

CONDITIONS: Adult
Keywords: Motor Learning; Feedback; Brain Function

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Performance Feedback (Experimental): Practice of a joystick based motor sequence task. Participants receive feedback on their response time to complete the trials in the practice block.
  Interventions: Behavioral: Motor Sequence Task
- Performance plus Positive Feedback (Experimental): Practice of a joystick based motor sequence task. Participants receive feedback on their response time to complete the trials in the practice block plus positive social comparative feedback.
  Interventions: Behavioral: Motor Sequence Task

INTERVENTIONS:
Behavioral: Motor Sequence Task — Participants will be seated at a laptop with the right hand on a standard joystick. The movement of the joystick will move a cursor on the computer screen. Targets will appear on the laptop screen as a circle in one of twelve spatially distinct locations. The learner must move the joystick "cursor" to inside the target before the next target will appear.

SUMMARY:
Feedback delivered during motor practice can help promote motor skill learning, enhance confidence, and alter brain connectivity. However, the optimal way to provide feedback to promote learning, confidence and brain connectivity is unknown. This project will study how the feedback that is provided during practice of a movement skill can help people learn and build confidence and whether these correspond to changes in brain function. The investigators will measure motor skill performance, confidence, and resting state brain connectivity before and after a session of motor practice.

DETAILED DESCRIPTION:
Positive social comparative feedback, which indicate to the learner that they are performing above average, is one way to enhance a learner's expectancies about future performance. Expectancies include the learners' perceived competence about their ability to perform the task, expectations about task outcome (success or failure), and predictions of extrinsic reward or positive experiences related to performance. Positive feedback during motor practice enhances expectancies, which is hypothesized to be rewarding to the learner, leading to better skill performance and learning. Reward is a powerful shaper of behavior. However, while social comparative feedback supports motor skill learning, it is unclear whether positive social comparative feedback induces a response in the dopamine reward network. Therefore, the purpose of this study is to determine the effects of social comparative feedback during motor practice on the functional connectivity of the reward neural network. The study aims to recruit 40 participants who will be randomized into 1 of 2 feedback groups (performance feedback or performance plus positive feedback). Participants will practice a motor sequence task on a single day and then return for retention performance testing about 24 hours later. Measures of brain function and brain structure will be collected before and after practice on day 1. Changes in performance (response time to complete a sequence) and self-efficacy will be measured from baseline to 24 hours later at retention. Changes in brain functional connectivity over practice on day 1 will be assessed in the reward network and the motor network.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 40 years
* Right-hand dominant

Exclusion Criteria:

* Medical diagnosis or medication that affects dopamine (e.g. dopamine reuptake inhibitors)
* Musculoskeletal issues that limit upper extremity movement
* Contraindications for magnetic resonance imaging (MRI)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-01-10 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Response Time | Change from baseline to retention at 24 hours
  Time to complete one sequence
Task Confidence | Change from baseline to retention at 24 hours
  Self-reported confidence in ability to complete a sequence in a given time on a scale of 0 to 10 with a 10 equating to higher confidence
Brain Connectivity | Change from baseline to immediately after practice
  Resting state connectivity between pairs of brain regions

SECONDARY OUTCOMES:
Peak Velocity | Change from baseline to retention at 24 hours
  Average speed to capture a target within a sequence
Total Path Distance | Change from baseline to retention at 24 hours
  Total distance traveled to complete one sequence
Time to Peak Velocity | Change from baseline to retention at 24 hours
  Mean time to peak velocity for movement to a target within a sequence
Perceived Competence | Change from baseline to retention at 24 hours
  Mean score on the Perceived Competence subscale of the Intrinsic Motivation Inventory where each item ranges from 0 to 7 with a higher value equating to higher competence
Perceived Interest/Enjoyment | Change from baseline to retention at 24 hours
  Mean score on the Interest/Enjoyment subscale of the Intrinsic Motivation Inventory where each item ranges from 0 to 7 with a higher value equating to higher enjoyment
Positive Affect | Change from baseline to retention at 24 hours
  Total score for general positive affect on the Positive and Negative Affect Scale with a range from 10 to 50 with higher scores equating to higher positive affect
Peak Velocity | Change from baseline to immediately after practice
  Average speed to capture a target within a sequence
Total Path Distance | Change from baseline to immediately after practice
  Total distance traveled to complete one sequence
Time to Peak Velocity | Change from baseline to immediately after practice
  Mean time to peak velocity for movement to a target within a sequence
Perceived Competence | Change from baseline to immediately after practice
  Mean score on the Perceived Competence subscale of the Intrinsic Motivation Inventory where each item ranges from 0 to 7 with a higher value equating to higher competence
Perceived Interest/Enjoyment | Change from baseline to immediately after practice
  Mean score on the Interest/Enjoyment subscale of the Intrinsic Motivation Inventory where each item ranges from 0 to 7 with a higher value equating to higher enjoyment
Positive Affect | Change from baseline to immediately after practice
  Total score for general positive affect on the Positive and Negative Affect Scale with a range from 10 to 50 with higher scores equating to higher positive affect
Response Time | Change from baseline to immediately after practice
  Time to complete one sequence
Task Confidence | Change from baseline to immediately after practice
  Self-reported confidence in ability to complete a sequence in a given time on a scale of 0 to 10 with a 10 equating to higher confidence
Brain Structure | Baseline assessment
  Structural integrity of white matter pathways in the brain

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available per reasonable request to the principal investigator 1 year after study completion.
Supporting Information: Study Protocol
Time Frame: 1 year after study completion